CLINICAL TRIAL: NCT02611180
Title: Analysis of Dendritic Cells in Patients With Acute or Chronic Skin Graft Versus Host Disease
Brief Title: Dendritic Cells in Patients With Acute or Chronic Skin Graft Versus Host Disease
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201405065
Record Dates: First submitted 2015-11-12; First posted 2015-11-20 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Acute Graft-versus-host Disease; Acute GVHD; Chronic Graft-versus-host Disease; Chronic GVHD
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin samples and blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm 1: Acute skin GVHD: * When clinically indicated, patients will undergo a skin biopsy to confirm a suspected diagnosis of acute or chronic GVHD, or to assess the status of their previously diagnosed acute or chronic GVHD. After the necessary samples are obtained for optimal medical care of the patient, two 6 mm punch biopsies (or four 4 mm punch biopsies) will be performed for research purposes, one (or two) of the affected area and one (or two) of a non-affected area (normal skin).
  * Patients who have clinical resolution of their acute or chronic GVHD will undergo one additional 6 mm punch biopsy (or two additional 4 mm punch biopsies) of the previously affected area. This additional biopsy should occur within 10 cm of the previous affected area sample.
  * With each skin biopsy, peripheral blood will be obtained by venipuncture or cannulation of an indwelling venous access device.
  * Two optional skin biopsies. One on day 5-7 of treatment and one on day 28 from the start of treatment.
  Interventions: Procedure: Skin punch biopsy; Procedure: Peripheral blood draw
- Arm 2: Chronic skin GVHD: * When clinically indicated, patients will undergo a skin biopsy to confirm a suspected diagnosis of acute or chronic GVHD, or to assess the status of their previously diagnosed acute or chronic GVHD. After the necessary samples are obtained for optimal medical care of the patient, two 6 mm punch biopsies (or four 4 mm punch biopsies) will be performed for research purposes, one (or two) of the affected area and one (or two) of a non-affected area (normal skin).
  * Patients who have clinical resolution of their acute or chronic GVHD will undergo one additional 6 mm punch biopsy (or two additional 4 mm punch biopsies) of the previously affected area. This additional biopsy should occur within 10 cm of the previous affected area sample.
  * With each skin biopsy, peripheral blood will be obtained by venipuncture or cannulation of an indwelling venous access device.
  * Two optional skin biopsies. One on day 5-7 of treatment and one on day 28 from the start of treatment.
  Interventions: Procedure: Skin punch biopsy; Procedure: Peripheral blood draw

INTERVENTIONS:
Procedure: Skin punch biopsy
Procedure: Peripheral blood draw

SUMMARY:
Dendritic cells (DCs) serve as sentries for the immune system. DCs recognize foreign compounds (antigens) in the body, which they internalize and process. When DCs uptake foreign antigens, they migrate to secondary lymphoid organs, where the processed antigens are presented to T cells.

Various DC subsets with unique cell lineages, surface protein markers, and tissue localization determinants have been identified. For example, Langerhans cells (LCs) and interstitial dendritic cells (intDCs) are DCs found in stratified epithelia, such as the skin. Though both are expressed in the skin, they differ with respect to their origin and surface protein content and can activate distinct types of immune responses. They may also have different specificities for the capture of antigens and presentation to circulating T cells.

To date, it is unknown what role, if any, the different DC populations that reside or repopulate in the skin play in the development and progression of skin graft-versus-host disease (GVHD) following bone marrow transplant.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at enrollment
* Willing and able to sign the informed consent
* Current diagnosis/suspected diagnosis of acute skin GVHD OR Current diagnosis/suspected diagnosis of chronic skin GVHD

Exclusion Criteria:

* Known infection with Hepatitis B or C, HTLV, or HIV
* Pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with current or suspected acute or chronic GVHD of the skin
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-04-30 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Dendritic cell characteristics | Up to 2 years
  * Both GVHD affected and unaffected skin sections will be analyzed by immunostaining and the types of cells and strains of skin microbiota present will be analyzed
  * The different isolated DCs will be activated by different stimuli and will be characterized by gene (DNA, RNA sequencing or arrays) and multicolor flow cytometry analysis.
Antigen specific lymphocyte subset characteristics | Up to 2 years
  * Both GVHD affected and unaffected skin sections will be analyzed by immunostaining and the types of cells and strains of skin microbiota present will be analyzed
  * CD4+ and CD8+ T cells or other lymphocyte populations will be isolated from peripheral blood by fluorescence activated cell sorting. The DC subsets purified from the skin tissue will be used to stimulate these T cell populations. This will be followed by thorough characterization of the charged T cell populations by a variety of methods. These will include assays to measure proliferation, gene array analysis cytokine secretion and other functions of the charged T cells.
Genes and skin microbiota that correlate with dendritic cell function | Up to 2 years
Potential treatment targets as measured by deep sequencing or microarray analysis | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Eynav Klechevsky, Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu